CLINICAL TRIAL: NCT03849859
Title: A Prospective Randomized Trial Comparing Single Plastic Stent Versus Multiple Plastic Stents in Inoperable Malignant Distal Bile Duct Obstruction.
Brief Title: Single Versus Multiple Plastic Stents in Malignant Distal Bile Duct Obstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of difficulty in completing the study as originally planned and loss of extra-funding.
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Nisa Netinatsunton, Principal Investigator, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC.61-096-21-1
Record Dates: First submitted 2019-02-13; First posted 2019-02-21 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2019-02

CONDITIONS: Plastic Stent Occlusion
Keywords: Plastic stent; Endoscopic Retrograde Cholangiopancreatography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single plastic stent (Active Comparator): Deployment of single plastic stent
  Interventions: Device: Single plastic stent
- Multiple plastic stents (Active Comparator): Deployment of multiple plastic stent
  Interventions: Device: Multiple plastic stents

INTERVENTIONS:
Device: Single plastic stent — Deployment of single plastic stent
  Arms: Single plastic stent
Device: Multiple plastic stents — Deployment of multiple plastic stents
  Arms: Multiple plastic stents

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) with biliary stent placement is crucial for palliative treatment in patients with malignant bile duct obstruction who cannot perform surgery due to advanced diseases or associated comorbidities. Stent patency is challenge in ERCP. Self expanding metallic stents (SEMS) have a longer duration of patency and fewer of recurrence occlusion of stent when compared with plastic stent (PS). However, the cost of MS is more expensive than PS about 4 times. Therefore, many patients cannot afford the MS due to their economic status. Data regarding the efficacy and safety of multiple PS compared with single PS for the palliative treatment in unresectable malignant distal bile duct obstruction are limited.

DETAILED DESCRIPTION:
The aim of the current study is to compare the cumulative stent patency of multiple PS and single plastic stent and the clinical success rate as a primary objective, investigate the technical success rate, procedure time incident of overall adverse events including stent dysfunction and overall procedure related mortality as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

In-operable distal malignant bile duct obstruction Age>18

Exclusion Criteria:

Pregnancy ECOG 3-4 Can not correct coagulopathy Contraindicate for ERCP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Cumulative stent patency | From the date of randomization though the study completion, assessed up to 1 year.
  Proportion of patients with documented stent dysfunction
Clinical success rate | Four weeks after randomization
  Proportion of patients with total bilirubin level declining > 50 % of the initial value

SECONDARY OUTCOMES:
Overall adverse events | From the date of randomization until the date of documented adverse events, assessed up to 1 month.
  Proportion of patients develop adverse events associated procedure included pancreatitis, cholangitis, hemorrhage.
Overall patient survival | From the date of randomization until the date of death from any cause, assessed up to 12 months.
  Proportion of patients who die from any causes.
Procedure relate death | From the date of randomization until the date of death from procedure within 7 days
  Proportion of patients who die from complications related procedure.
Technical success rate | From the date of randomization until the last stent deploy, assessed up to 1 day.
  Proportion of patient who successful underwent stent placement.

CONTACTS AND LOCATIONS:
Overall Officials: Ni Netinatsunton, M.D., Principal Investigator — NKC Institute of Gastroenterology and Hepatology.
Locations (2):
- Thailand (2):
  - NKC Institue of Gastroenterology and Hepatology, Prince of Songkla University, Hat Yai, Changwat Songkhla
  - NKC Institues of Gastroenterology and Hepatology, Prince of Songkla University, Hat Yai, Changwat Songkhla

IPD SHARING:
Plan to Share IPD: No